CLINICAL TRIAL: NCT06728423
Title: SmartGuard vs Temp Target in Patients With Type 1 Diabetes Users AHCL in Anaerobic Exercise
Brief Title: Comparison of SmartGuard vs Temp Target in Patients With Type 1 Diabetes Users of Advanced Hybrid Closed Loop System (AHCL) in Anaerobic Physical Activity.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FM-CIE-1333-23
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D); Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Temporary Target (Other): Temporary target during an anaerobic training session
  Interventions: Other: Temporary target during an anaerobic training session
- SmartGuard (Other): SmartGuard during an anaerobic training session
  Interventions: Other: SmartGuard during an anaerobic training session

INTERVENTIONS:
Other: Temporary target during an anaerobic training session — Temporary target during an anaerobic training session
  Arms: Temporary Target
Other: SmartGuard during an anaerobic training session — SmartGuard during an anaerobic training session
  Arms: SmartGuard

SUMMARY:
Patients meeting the inclusion criteria will be identified. An informed consent form will be completed. Clinical data and baseline CGM will be collected at this appointment. During the session, an attempt will be made to establish a physical activity classification (PA0: inactive, PA1: 1-2 times per week, and PA2: more than twice per week) to determine if the patient is physically active, which is defined as at least 60 minutes of physical activity per week during the past 6 months. In addition, the patient will be asked whether or not they perform strength exercises and how regularly they do so. At the end of the first visit, they will be randomized by an electronically generated numerical sequence using the Randomizer for Clinical Trial Lite application. The patient will be scheduled to attend a supervised exercise session at the Pontificia Universidad Javeriana Sports Training Center.

Participants will have a blood glucose test prior to beginning physical activity. The target for starting exercise is 126-180 mg/dl. If the patient has a value less than 90 mg/dl, 20 grams of carbohydrates will be given; if the value is between 90-126 mg/dl, 10 grams will be given (above the investigators said that for anaerobics it could be from 90 mg/dl). If the value is higher than 200 mg/dl, the correction with rapid insulin is calculated according to your usual management. A new glucose test is performed 15 minutes later to confirm that the patient is within the target range. If the patient is within the target range, exercise is performed. If the reading remains above 200, the exercise session is canceled.

All participants are in SmartGuard mode on the Minimed 780G system. In the control group, the time target is activated 60 minutes before the activity and turned off 15 minutes after the end of the exercise. Participants randomized to SmartGuard will have no changes in device programming. Glucose measurements will be taken at the beginning and end of the exercise session. In addition, a Hooper Index will be calculated to standardize the patient's rest and recovery prior to the session. The strength training session will begin with a brief 15-minute warm-up emphasizing joint flexibility. The workout will consist of 3 sets of 10 repetitions of the following exercises: leg press, chest press, seated row. The estimated weight at which the exercises will be performed will be 60-80% of the 1-RM calculated for each patient. There will be a 90 second timed rest between each set of exercises. The total duration of the training will be 45 minutes. The strength training session begins with a short 15-minute warm-up focusing on joint flexibility. The workout consists of 3 sets of 10 repetitions of the following exercises: leg press, chest press, seated row. The estimated weight at which the exercises are performed is 60-80% of the 1-RM calculated for each patient. A timed rest of 90 seconds will be provided between each set of exercises. The total duration of the training will be 45 minutes. The parameter used to monitor intensity will correspond to the Borg scale measurement and heart rate monitoring. For each participant, the anthropometric variables will be entered into the application in order to perform the exact calculation of the target maximum heart rate (HR) percentage. The activity begins with a 5-minute warm-up at low intensity (55-65% of maximum HR, Borg 9-11), then 35 minutes at moderate intensity (70-80% of maximum HR, Borg 12-13), and ends with a 5-minute cool-down (maximum HR less than 55%). Alarms are set on the device to maintain the desired intensity. Glucose testing is performed at the beginning and end of the activity.

A 14-day washout period will be carried out, after which the group of patients initially assigned to temporary target activation will perform the same exercise in SmartGuard mode; likewise, the group initially assigned to SmartGuard will do so under temporary target mode. For this second session, the same procedure and recommendations already mentioned will be carried out.

CGM data will be collected through integrated continuous glucose monitoring, which downloads the information to the Carelink portal and is accessed online.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes ≥ 1 year ago
* AHCL users (Minimed 780G) with integrated continuous glucose monitoring
* Use of the device for at least the last 3 months
* Physically active (PA≥1): At least one weekly physical exercise session in the last 6 months.

Exclusion Criteria:

* Pregnancy
* Physical or mental inability to exercise
* Contraindication to performing Valsalva maneuvers
* History of osteoarticular disease that prevents exercise
* History of tendinopathies that cause pain or limitation
* History of coronary artery disease
* Diabetic ketoacidosis or severe hypoglycemia in the last month
* Evidence of autonomic failure (Unnoticed hypoglycemia given by Clarke 3 or more points Appendix 1) I am concerned because now that I am on a pump, this indication is common as support for the insulin pump.
* Use of beta-blockers or glucocorticoids
* Peripheral arterial disease
* Severe proliferative diabetic retinopathy or non-proliferative diabetic retinopathy
* Severe peripheral neuropathy
* Stage 5 chronic kidney disease on renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Time in range | 30 days
  To compare the difference in glycemic control (TIR and GMI) and safety (TBR and hypoglycemic events) of time-based target activation versus SmartGuard mode in type 1 diabetic patients using the MiniMed 780G during anaerobic exercise.

SECONDARY OUTCOMES:
Hypoglycemia <54 mg/dl | 30 days
  Determination and comparison of rates of clinically significant hypoglycemia
Time in range according phases | 30 days
  Compare the percentage of time in range in the immediate, early, and late phases of the strength exercise.
Time Below Range <70 mg/dl. | 30 days
  Compare the percentage of time below range in the immediate, early, and late phases of the strength exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Ignacio., Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
For research purposes, the data will be made available to the reader upon request.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: For research purposes, the data will be made available to the reader upon request.